CLINICAL TRIAL: NCT04311879
Title: Efficiency of Soft Tissue Diode Laser Application on Healing of Periapical Tissues (A Randomized Clinical Trial)
Brief Title: Efficiency of Soft Tissue Diode Laser Application on Healing of Periapical Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hend Hamdy Ismail, PhD candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: END 16-14D
Record Dates: First submitted 2020-03-07; First posted 2020-03-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Periapical Diseases
Keywords: Diode laser; low level laser therapy; CBCT
MeSH Terms: conditions — Periapical Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft tissue laser Diode laser application (Experimental): Endodontically treated teeth by virtue of a dental applicator positioned at a right angle to the mucosa at the level of the apices. Application of the laser probe was applied to both the buccal and lingual mucosae overlying the apices of the target tooth. Total exposure time for each tooth was 60 seconds (a dose = 70 j/cm2 for analgesia) The laser unit used in this study used was a diode laser (Lite Medics 1.00Watt serial number 148 Ver.SwvM. 150VS108VT.100) of wavelength 980nm and Max power 15WCW Class IV Laser Product
  Interventions: Device: Soft tissue Diode laser application
- conventional root canal treatment (Placebo Comparator): Placebo : conventional root canal conventional root canal treatment with irrigation of sodium hypochlorite 2.5% with mock laser intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Soft tissue Diode laser application — post-operative soft tissue diode laser application
  Other Names: Low laser therapy
  Arms: Soft tissue laser Diode laser application
Other: Placebo — mock diode laser application
  Arms: conventional root canal treatment

SUMMARY:
Study is a Randomized clinical trial conducted at Endodontic department- Ain Shams university Cairo. Egypt. 24 eligible patients were selected and included in the study to compare healing ability of soft tissue diode laser application versus conventional root canal treatment using CBCT

DETAILED DESCRIPTION:
Sample size is 24 24 Patients were randomly distributed in 2 groups , one group of patients received soft tissue laser therapy after root canal treatment and the other group received no treatment just conventional RCT. • Patients were equally divided into 2 groups (n=12 in each group ) The study in a Single blinded RCT , Numbers for patients will be generated and distributed randomly in a table on an Excel sheet, and in front of each number either a letter (C) for control or (I) for intervention will be typed After patients were selected in the study they will be asked to fill in a consent form , that states that they are part of a clinical trial and that they may or may not have a laser session following root canal treatment Group A Soft tissue laser application : Endodontically treated teeth were targeted by virtue of a dental applicator positioned at a right angle to the mucosa at the level of the apices. Application of the laser probe were applied to both the buccal and lingual mucosae overlying the apices of the target tooth. Total exposure time for each tooth was 60 seconds (a dose = 70 j/cm2 for analgesia) by the co-investigator The laser unit used in this study will be a diode laser (Lite Medics 1.00 Watt serial number 148 Ver.SwvM. 150VS108VT.100) of wavelength 980nm and Max power 15 WCW Class IV Laser Product ) in continuous wave mode Group B : Placebo : conventional root canal treatment : mock laser intervention A CBCT was taken preoperative and after 12 month postoperative, both linear and volumetric measurements were calculated

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age between 18-50 years
* Medically free patients.
* Patients suffering from acute or chronic infection with symptomatic apical periodontitis with Necrotic pulp
* Preoperative Pain
* Sensitivity to percussion
* Periapical radiographic X-ray showing periapical lesion with no gutta percha in canal
* Occlusal contact with opposing teeth

Exclusion Criteria:

* Pregnant females.
* Patients having a significant systemic disorder or history of drug abuse
* Patients who had administrated analgesics or antibiotics during the last 12 hours preoperatively.
* Patients having bruxism or clenching
* Teeth having:

  * No occlusal contact
  * No sensitivity to percussion
  * Greater than grade I mobility.
  * Pocket depth greater than 5mm.
  * No possible restorability
  * Procedural errors
  * Previous Root canal treatment
  * Open apex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Assess post-operative healing in a period of 12 month when using Soft tissue diode laser application post-operative using CBCT | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maram Obeid, PhD, Study Director — AinShams University; Ehab Hassanien, PhD, Study Chair — Ainshams University
Locations (1):
- Endodontic department - Faculty of Dentistry Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No